CLINICAL TRIAL: NCT01587755
Title: Optimising Outpatient Care in Mild to Moderate Psoriasis by a Newly Developed 'Topical Treatment Optimising Programme' - an International Study Using Daivobet®/Dovobet® Gel
Brief Title: Optimising Outpatient Care in Mild to Moderate Psoriasis (PSO-TOP)
Acronym: PSO-TOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kristian Reich, MD (Individual)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor-Investigator, Kristian Reich, MD, Kristian Reich, MD, Reich, Kristian, M.D.
Organization: Reich, Kristian, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 055-006
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Mild to Moderate Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Treatment Optimizing Program (Other): Optimized care
  Interventions: Other: TTOP
- non-Topical Treatment Optimizing Program (Other): Standard care
  Interventions: Other: non-TTOP

INTERVENTIONS:
Other: TTOP — Patient is taken care of in an intensified, optimised manner
  Arms: Topical Treatment Optimizing Program
Other: non-TTOP — Standard medical care
  Arms: non-Topical Treatment Optimizing Program

SUMMARY:
A Topical Treatment Optimisation Programme (TTOP) has been developed by the sponsor together with Patient Boards and an Expert Advisory Board to overcome non-adherence problems.

DETAILED DESCRIPTION:
A Topical Treatment Optimisation Programme (TTOP) has been developed by the sponsor together with Patient Boards and an Expert Advisory Board. This tool is created to address patients' non-adherence in topical therapy and the resulting underperformance of such treatments in controlling psoriatic disease. The study addresses the effect of the relationship between the patient and the health care professional, one of the important factors that can affect treatment adherence and therapeutic efficacy. The TTOP will be compared to standardised regular care (called 'non-TTOP'). It is intended to clinically show the importance of an optimised contact between the patient and health care professional.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged at least 18 years
* Mild to moderate active plaque psoriasis with PGA ≥ 2 on the 7-point scale by Langley and Ellis and a Body Surface Area (BSA) of ≤ 10%
* Topical psoriasis treatment with coal or tar preparations, tazarotene, steroids, or vitamin D analogues, or combinations of steroids and vitamin D analogues (except gel combination products containing 50 micrograms calcipotriol/0.5mg betamethasone/g) or dithranol and its combination preparations over the last 8 weeks prior to Visit 1 (week 0)
* Written informed consent to participate in the study has been given prior to any study related procedures

Exclusion Criteria:

* Severe renal insufficiency
* Severe hepatic disorders
* Known hyper calcaemia
* Erythrodermic, exfoliative, pustular or guttate psoriasis
* Facial or genital psoriasis
* Fulfilment of at least one contraindication according to the Summary of Product Characteristics of Daivobet®/Dovobet® Gel
* Pregnant and/or breast-feeding women
* Hypersensitivity to the active substances or to any of the excipients
* Suspected non-compliance with the clinical study procedures
* Current participation in another clinical study
* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to Visit 1 (week 0):

  * etanercept - within 4 weeks prior to Visit 1 (week 0)
  * adalimumab, alefacept, infliximab - within 2 months prior to Visit 1 (week 0)
  * ustekinumab - within 4 months prior to Visit 1 (week 0)
  * experimental products - within 4 weeks/5 half-lives (whichever is longer) prior to Visit 1 (week 0)
* Phototherapy within the following time periods prior to Visit 1 (week 0):

  * PUVA - within 4 weeks prior to Visit 1 (week 0)
  * UV-B - within 2 weeks prior to Visit 1 (week 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1852 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Physician Global Assessment (PGA) | Up to 64 weeks; primary outcome assessed at week 8 after treatment start
  PGA (Physician Global Assessment) will be assessed at all study visits. For week 8, the rate of patients with a PGA (as defined by Langley and Ellis 2004) of 0 or 1 will be calculated. This is the primary study parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Reich, MD Prof., Principal Investigator
Locations (93):
- Denmark (4):
  - Herning
  - Hobro
  - Roskilde
  - Vejle
- France (14):
  - Angers
  - Auxerre
  - Brest
  - Lille
  - Limeil-Brévannes
  - Marseille
  - Martigues
  - Paris
  - Poitiers
  - Saint-Germain-en-Laye
  - Saint-Mandé
  - Saint-Priest-en-Jarez
  - Tours
  - Vienne
- Germany (21):
  - Bad Bentheim
  - Berlin
  - Biberach
  - Blaubeuren Abbey
  - Bochum
  - Buchholz
  - Cologne
  - Dessau
  - Frankfurt
  - Friedrichshafen
  - Gilching
  - Hamburg
  - Hanover
  - Kiel
  - Mahlow
  - Osnabrück
  - Pinneberg
  - Selters
  - Weißenfels
  - Wolfenbüttel
  - Wuppertal
- Italy (14):
  - Brescia
  - Catania
  - Genova
  - Lucca
  - L’Aquila
  - Messina
  - Padua
  - Palermo
  - Parma
  - Pavia
  - Perugia
  - Rome
  - Trapani
  - Verona
- Netherlands (5):
  - Amsterdam
  - Geldrop
  - Maastricht
  - Nijmegen
  - Rotterdam
- Spain (9):
  - Alicante
  - Barcelona
  - Fuenlabrada (Madrid)
  - Getafe (Madrid)
  - Madrid
  - Palma de Mallorca
  - Tarragona
  - Valencia
  - Zaragoza
- Sweden (6):
  - Eskilstuna
  - Gothenburg
  - Kristianstad
  - Linköping
  - Örebrö
  - Uppsala
- United Kingdom (20):
  - Bexhill-on-Sea
  - Bradford
  - Burbage
  - Canterbury
  - Cheshire
  - Chesterfield
  - Coventry
  - Darwen
  - East Sussex
  - London
  - Manchester
  - Merseyside
  - Middlesex
  - Nantwich
  - Nuneaton
  - Oldham
  - Royal Leamington Spa
  - Royal Tunbridge Wells
  - Warwickshire
  - West Sussex

REFERENCES:
- [Background] Reich K, Zschocke I, Bachelez H, de Jong EM, Gisondi P, Puig L, Warren RB, Mrowietz U; TTOP study group. Efficacy of a fixed combination of calcipotriol/betamethasone dipropionate topical gel in adult patients with mild to moderate psoriasis: blinded interim analysis of a phase IV, multicenter, randomized, controlled, prospective study. J Eur Acad Dermatol Venereol. 2015 Jun;29(6):1156-63. doi: 10.1111/jdv.12774. Epub 2014 Oct 26. PMID 25346093
- [Background] Reich K, Mrowietz U, Karakasili E, Zschocke I. Development of an adherence-enhancing intervention in topical treatment termed the topical treatment optimization program (TTOP). Arch Dermatol Res. 2014 Sep;306(7):667-76. doi: 10.1007/s00403-014-1475-5. Epub 2014 Jun 4. PMID 24895177
- [Background] Zschocke I, Mrowietz U, Lotzin A, Karakasili E, Reich K. Assessing adherence factors in patients under topical treatment: development of the Topical Therapy Adherence Questionnaire (TTAQ). Arch Dermatol Res. 2014 Apr;306(3):287-97. doi: 10.1007/s00403-014-1446-x. Epub 2014 Feb 8. PMID 24509981
- [Derived] Reich K, Zschocke I, Bachelez H, de Jong EMGJ, Gisondi P, Puig L, Warren RB, Ortland C, Mrowietz U; PSO-TOP study group. A Topical Treatment Optimization Programme (TTOP) improves clinical outcome for calcipotriol/betamethasone gel in psoriasis: results of a 64-week multinational randomized phase IV study in 1790 patients (PSO-TOP). Br J Dermatol. 2017 Jul;177(1):197-205. doi: 10.1111/bjd.15466. Epub 2017 Jun 6. PMID 28301043